CLINICAL TRIAL: NCT03328130
Title: Safety and Efficacy of a Unilateral Subretinal Administration of HORA-PDE6B in Patients With Retinitis Pigmentosa Harbouring Mutations in the PDE6B Gene Leading to a Defect in PDE6ß Expression
Brief Title: Safety and Efficacy Study in Patients With Retinitis Pigmentosa Due to Mutations in PDE6B Gene
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of financing
Sponsor: eyeDNA Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HORA-PDE6B-001; 2016-001429-16 (EudraCT Number)
Record Dates: First submitted 2017-10-05; First posted 2017-11-01 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Retinitis Pigmentosa
Keywords: Adeno-associated virus; AAV; Retinitis Pigmentosa; PDE6B; Gene Therapy; Gene Transfer; Retinal Dystrophy; Eye Diseases; Vision Disorders; Eye Diseases, Hereditary; Retinal Diseases; Retinal Degeneration
MeSH Terms: conditions — Retinitis Pigmentosa; Retinal Dystrophies; Eye Diseases; Vision Disorders; Eye Diseases, Hereditary; Retinal Diseases; Retinal Degeneration

STUDY DESIGN:
Intervention Model Description: Five successive cohorts separated by DSMC assessments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort 1 - Low Dose (Experimental): Biological: AAV2/5-hPDE6B Unilateral (one eye), subretinal, administration of the lowest dose. Dose-escalation will be performed after DSMC assessment.
  Interventions: Biological: AAV2/5-hPDE6B
- Cohort 2a - Medium Dose (Experimental): Biological: AAV2/5-hPDE6B Unilateral (one eye), subretinal, administration of the medium dose. Confirmatory dose will be determined after DSMC assessment.
  Interventions: Biological: AAV2/5-hPDE6B
- Cohort 2b - High Dose (Experimental): Biological: AAV2/5-hPDE6B Unilateral (one eye), subretinal, administration of the highest dose. Confirmatory dose will be determined after DSMC assessment.
  Interventions: Biological: AAV2/5-hPDE6B
- Cohort 3 - High Dose (confirmatory cohort) (Experimental): Biological: AAV2/5-hPDE6B Unilateral (one eye), subretinal, administration of the confirmatory dose.
  Interventions: Biological: AAV2/5-hPDE6B
- Cohort 4 - High Dose - 13 years old or older population (Experimental): Biological: AAV2/5-hPDE6B Unilateral (one eye), subretinal, administration of the confirmatory dose.
  Interventions: Biological: AAV2/5-hPDE6B

INTERVENTIONS:
Biological: AAV2/5-hPDE6B — Subretinal administration in one eye

SUMMARY:
The study is a Phase I/II, monocentric, open-label, dose-ranging safety and efficacy gene therapy intervention by subretinal administration of AAV2/5-hPDE6B.

At least twelve patients 18 years of age or older, within four consecutive cohorts of patients, will be recruited.

Then at least four patients 13 years of age or older, within a fifth cohort, will be recruited.

DETAILED DESCRIPTION:
Retinitis pigmentosa (RP) is a disease where part of the eye (the retina) is degenerating over time. Patients initially present with night blindness, and later in life experience loss of central vision which leads to blindness. RP is a highly variable disorder with some patients developing symptomatic visual loss in childhood whereas others remain asymptomatic until mid-adulthood. There are no treatments available.

This study focuses on the form of RP caused by mutations (modifications) in the genetic information necessary to make the protein called rod cGMP phosphodiesterase 6 β subunit (or PDE6β). Clinical diagnosis is made by function tests of the eye and confirmed using a specific method called molecular testing to verify that the PDE6B gene is not correct.

This study uses a gene therapy vector inspired from an adeno-associated virus (AAV) called AAV2/5-hPDE6B. This vector intends to supply to the target cells the PDE6B therapeutic gene that is not functioning properly in the cell. The AAV parts of the gene therapy vector work as a vehicle to deliver the normal human PDE6B gene into the cells of the retina.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical and molecular diagnosis of retinitis pigmentosa caused by defect in PDE6B gene without other syndromic manifestations
* Aged above 13 years
* Ability to give informed consent

Key Exclusion Criteria:

* Previous ocular surgery or thermal laser within 6 months before the surgery
* Lens opacities or obscured ocular media upon recruitment such reliable evaluation or grading of the posterior segment cannot be performed
* Known serious allergies to the fluorescein dye used in angiography, to the mydriatic, steroidal and non-steroidal eye drops
* Participation in another clinical trial with an investigational agent
* Enrolled or being enrolled in another gene therapy clinical trial
* Active, extraocular infection requiring the prolonged or chronic use of antimicrobial agents
* Chronic medical conditions, cancer
* Abnormal laboratory values
* On immunosuppressive therapy

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of ocular and non-ocular adverse events | 1 year + 4 years follow-up

SECONDARY OUTCOMES:
Improvement in visual function | 1 year + 4 years follow-up
  Improvement in visual function as assessed by mobility test
Improvement in visual fields | 1 year + 4 years follow-up
  Improvement in visual fields as assessed by visual fields measurements
Improvement in visual function | 1 year + 4 years follow-up
  Improvement in visual function as assessed by reading speed
Improvement in Quality of Life | 1 year + 4 years follow-up
  Quality of life will be measured by Quality of Life questionnaire National Eye Institute Visual Function Questionnaire (NEI VFQ-25)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Ophtalmologique, CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Petit L, Lheriteau E, Weber M, Le Meur G, Deschamps JY, Provost N, Mendes-Madeira A, Libeau L, Guihal C, Colle MA, Moullier P, Rolling F. Restoration of vision in the pde6beta-deficient dog, a large animal model of rod-cone dystrophy. Mol Ther. 2012 Nov;20(11):2019-30. doi: 10.1038/mt.2012.134. Epub 2012 Jul 24. PMID 22828504
- [Result] Pichard V, Provost N, Mendes-Madeira A, Libeau L, Hulin P, Tshilenge KT, Biget M, Ameline B, Deschamps JY, Weber M, Le Meur G, Colle MA, Moullier P, Rolling F. AAV-mediated Gene Therapy Halts Retinal Degeneration in PDE6beta-deficient Dogs. Mol Ther. 2016 May;24(5):867-76. doi: 10.1038/mt.2016.37. Epub 2016 Feb 9. PMID 26857842
- [Derived] Palmowski-Wolfe A, Stingl K, Habibi I, Schorderet D, Tran HV. Novel PDE6B Mutation Presenting with Retinitis Pigmentosa - A Case Series of Three Patients. Klin Monbl Augenheilkd. 2019 Apr;236(4):562-567. doi: 10.1055/a-0811-5480. Epub 2019 Jan 15. PMID 30646425